CLINICAL TRIAL: NCT07295093
Title: Association Between Age at Menopause and Levels of Anxiety and Depression
Brief Title: Menopause Age and Anxiety-Depression
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Didem Eşkin Tanrıverdi, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-25-1981
Record Dates: First submitted 2025-12-04; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Menopause; Primary Ovarian Insufficiency (Poi); Anxiety; Depression; Menopausal Depression
Keywords: Menopause; Primary Ovarian Insufficiency (Poi); Anxiety; depression
MeSH Terms: conditions — Primary Ovarian Insufficiency; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Menopause group: Patients over 40 years of age who have undergone menopause and who visited our hospital's obstetrics and gynecology outpatient clinic for routine check-ups, without any additional diseases or complaints.
  Interventions: Other: Beck Anxıety Inventory (BAI); Other: State-Trait Anxiety Scale (STAI) 1-2
- Primary ovarian insufficiency (POI) group: Patients who experienced menopause before the age of 40 and who visited our hospital's obstetrics and gynecology outpatient clinic for routine check-ups, without any additional diseases or complaints.
  Interventions: Other: Beck Anxıety Inventory (BAI); Other: State-Trait Anxiety Scale (STAI) 1-2

INTERVENTIONS:
Other: Beck Anxıety Inventory (BAI) — Beck Anxıety Inventory (BAI) Description: The scale will be self-administered and completed by the patient during the routine outpatient clinic visit.
  Other Names: State-Trait Anxiety Scale (STAI) 1-2
Other: State-Trait Anxiety Scale (STAI) 1-2 — State-Trait Anxiety Scale (STAI) 1-2 Description: The scale will be self-administered and completed by the patient during the routine outpatient clinic visit.

SUMMARY:
Menopause is defined as the permanent cessation of menstrual cycles due to ovarian follicle depletion, typically occurring after age 50, and is associated with decreased estrogen levels. Primary ovarian insufficiency (POI) involves early ovarian dysfunction before age 40, with infertility as a key concern. Both menopause and POI may contribute to psychological symptoms, including anxiety and depression, influenced by sociodemographic and health factors. While literature reports anxiety in middle-aged women, data on its association with menopausal timing are limited. This study aims to compare women with POI and those undergoing natural menopause after age 40, assessing the relationship between age at menopause, anxiety, and depression, as well as the impact of fertility expectations on psychological well-being in POI patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women over 24 years of age who visited our hospital for routine outpatient check-ups, had been diagnosed with menopause, and had no history of psychiatric disorders before menopause.

Exclusion Criteria:

* Cardiovascular diseases including hypertension
* Type 1 or type 2 diabetes mellitus
* Morbid obesity
* Primary adrenal insufficiency
* Uterine fibroids
* Thyroid dysfunctions including Hashimoto thyroiditis and Grave's disease
* Hepatic dysfunctions
* Renal insufficiency
* Genetic disorders in chromosome constitution or karyotype analysis including monosomy X, trisomy X and gene mutations as BMP15, FMR I, POFIB, and GDF9
* Neurologic diseases
* Psychiatric disorders
* Autoimmune diseases or syndromes including Addison's disease, autoimmune syndromes, scleroderma, Sjogren's syndrome, myasthenia gravis, inflammatory bowel diseases, multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus and familial Mediterranean fever
* History of any malignancy
* History of exposure to chemotherapeutic agents or radiotherapy
* Individuals with a history of chronic or regular medication use that could cause anxiety or depression symptoms
* Individuals with a personal history of psychiatric disorders
* Individuals with a history of depression in the past 6 months.

Min Age: 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible: Female participants only. This study specifically includes women who have undergone menopause, as well as women diagnosed with primary ovarian insufficiency (POI).
  Not Eligible: Male participants and individuals who do not identify as female.
Study Population: A total of 136 participants were included in the study, of whom 83 were in the menopause group and 53 in the primary ovarian insufficiency group.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Beck Anxıety Inventory (BAI), Anxiety level | Baseline (single assessment at enrollment during routine clinic visit).
  Anxiety severity measured by the Beck Anxiety Inventory (BAI) during routine clinic visit.
State-Trait Anxiety Scale (STAI) 1-2, Anxiety level | Baseline (single assessment at enrollment during routine clinic visit).
  Anxiety severity measured by the State-Trait Anxiety Inventory (STAI) forms 1 and 2 during routine clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Didem Eşkin Tanrıverdi, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Not Valid, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD are available which may be shared in necessary conditions.

REFERENCES:
- [Background] Bromberger JT, Meyer PM, Kravitz HM, Sommer B, Cordal A, Powell L, Ganz PA, Sutton-Tyrrell K. Psychologic distress and natural menopause: a multiethnic community study. Am J Public Health. 2001 Sep;91(9):1435-42. doi: 10.2105/ajph.91.9.1435. PMID 11527777
- [Background] Zollner YF, Acquadro C, Schaefer M. Literature review of instruments to assess health-related quality of life during and after menopause. Qual Life Res. 2005 Mar;14(2):309-27. doi: 10.1007/s11136-004-0688-z. PMID 15892422
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Bryant C, Judd FK, Hickey M. Anxiety during the menopausal transition: a systematic review. J Affect Disord. 2012 Jul;139(2):141-8. doi: 10.1016/j.jad.2011.06.055. Epub 2011 Jul 23. PMID 21783260
- [Background] Grigolon RB, Ceolin G, Deng Y, Bambokian A, Koning E, Fabe J, Lima M, Gerchman F, Soares CN, Brietzke E, Gomes FA. Effects of nutritional interventions on the severity of depressive and anxiety symptoms of women in the menopausal transition and menopause: a systematic review, meta-analysis, and meta-regression. Menopause. 2023 Jan 1;30(1):95-107. doi: 10.1097/GME.0000000000002098. Epub 2022 Nov 7. PMID 36576445